CLINICAL TRIAL: NCT07270809
Title: To Study the Clinical Course and Outcomes of Non-electively Hospitalised Patients of Chronic Liver Disease (CLD) With Hepatic or Extra-hepatic Predominant Organ Failure(s) at 6 Months.
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-CLD-66
Record Dates: First submitted 2025-04-02; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Liver Disease (CLD) With Hepatic Predominant Organ Failure
  Interventions: Other: No Intervention
- Chronic Liver Disease (CLD) With Extra-hepatic Predominant Organ Failure
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
Title - To study the clinical course and outcomes of non-electively hospitalised patients of chronic liver disease (CLD) with Hepatic or Extra-hepatic predominant organ failure(s) at 6 months.

Summary - ACLF is a condition where acute insult leading to worsening liver failure with or without extra-hepatic failure leads to a high short-term mortality. However, the presence of cirrhosis, prior decompensation, non-hepatic/systemic acute insult, organ failure and treatment are different in different part of the world. This is due to in-homogenous patient cohort. The current study was planned for all patients of CLD, who were non-electively hospitalized and were followed up for long-term to identify the differences in clinical course, acute insult, organ failure, therapy and outcome in relation to liver failure with or without extra-hepatic organic failure. In the study the laboratory, clinical parameters, inflammatory and regenerative markers will be evaluated as a marker of disease progression, reversal, recompensation or regression. This will enable us to differentiate the ACLF between east and west, guide us for defining the natural course of CLD with failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. CLD with or without cirrhosis with 1st or subsequent admissions for decompenasation and irrespective of any prior decompensation
3. Non-electively hospitalized

Exclusion Criteria:

1. HCC
2. NCPF/EHPVO
3. Pregnancy
4. Post-Liver transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Liver Disease with or without cirrhosis, non-electively hospitalized with decompensation, hepatic and/or extra-hepatic organ failure with/without prior decompensation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Death or liver transplant at 6 months follow up. | 6 months

SECONDARY OUTCOMES:
Recovery as per disease severity scores, i.e- decrease in MELD ≥5 and CTP ≥3 | 6 months
Organ dysfunction and organ failures | day 28, day 90, day 180

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided